CLINICAL TRIAL: NCT04840927
Title: An Open-Label, Single Center, Randomized, Pharmacoscintigraphic Study to Evaluate the Relative Bioavailability of E7386 Following Oral Administration of Targeted Release Tablets Compared to an E7386 Immediate Release Tablet in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability of E7386 Following Oral Administration of Targeted Release (TR) Tablets Compared to an E7386 Immediate Release (IR) Tablet in Healthy Adult Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Delay in availability of IMP
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E7386-E044-002; QSC203335 (Other: Quotient Sciences); 2020-005638-13 (EudraCT Number)
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: Relative Bioavailability; Pharmacoscintigraphic; Pharmacokinetic; E7386
MeSH Terms: interventions — E-7386

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: E7386 40 mg (Experimental): Participants will be randomized to one of the 3 treatment sequences:
  Treatment sequence 1: Participants will receive Regimen A on Day 1 of treatment period 1 then Regimen B on Day 1 of treatment period 2 then Regimen C on Day 1 of treatment period 3 and an optional Regimen D on Day 1 of an optional treatment period 4.
  Treatment sequence 2: Participants will receive Regimen B on Day 1 of treatment period 1 then Regimen C on Day 1 of treatment period 2 then Regimen A on Day 1 of treatment period 3 and an optional Regimen D on Day 1 of an optional treatment period 4.
  Treatment sequence 3: Participants will receive Regimen C on Day 1 of treatment period 1 then Regimen A on Day 1 of treatment period 2 then Regimen B on Day 1 of treatment period 3 and an optional Regimen D on Day 1 of an optional treatment period 4.
  A maximum wash out period of 10 days will be maintained between treatment periods 1, 2 and 3.
  Interventions: Drug: E7386
- Cohort 2: E7386 40 mg (Experimental): Participants will be randomized to one of the 3 treatment sequences:
  Treatment sequence 4: Participants will receive Regimen C on Day 1 of treatment period 1 then Regimen B on Day 1 of treatment period 2 then Regimen A on Day 1 of treatment period 3 and an optional Regimen D on Day 1 of an optional treatment period 4.
  Treatment sequence 5: Participants will receive Regimen A on Day 1 of treatment period 1 then Regimen C on Day 1 of treatment period 2 then Regimen B on Day 1 of treatment period 3 and an optional Regimen D on Day 1 of an optional treatment period 4.
  Treatment sequence 6: Participants will receive Regimen B on Day 1 of treatment period 1 then Regimen A on Day 1 of treatment period 2 then Regimen C on Day 1 of treatment period 3 and an optional Regimen D on Day 1 of an optional treatment period 4.
  A maximum wash out period of 10 days will be maintained between treatment periods 1, 2 and 3.
  Interventions: Drug: E7386

INTERVENTIONS:
Drug: E7386 — Regimen A: 40 milligram (mg) IR Oral Tablet.

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetic (PK) profile of E7386 following oral administration of E7386 enteric coated TR prototype tablet formulations (TR1, TR2 and optional TR3) and to evaluate the relative bioavailability of E7386 TR tablets compared to E7386 IR reference tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female (women of nonchildbearing potential [WNCBP]) aged greater than or equal to (>=) 30 years and less than or equal to (<=) 55 years old inclusive at the time of signing informed consent
2. Body Mass Index (BMI) >=18.0 and <=30.0 kilogram per square meter (kg/m^2) as measured at screening
3. Participants must demonstrate their ability to swallow an empty size 000 capsule (26.1*9.91 millimeter [mm]) at screening and must be willing and able to take the SmartPill^Trade Mark (TM) (27*12 mm)
4. Provide written informed consent
5. Willing and able to comply with all aspects of the protocol
6. Participant must have regular bowel movements (that is, average stool production of >=1 and <=3 stools per day)
7. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 millisieverts (mSv) in the last 12 months or 10 mSv in the last 5 years prior to Day -1 of Period 1. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
2. Male participants with pregnant or breastfeeding partners
3. Males who are unwilling to follow the contraception rules of the study for up to 92 days after last dose of the study drug
4. Females who are of childbearing potential or breastfeeding or pregnant at screening or admission/predose (as documented by a positive beta-human chorionic gonadotropin [or human chorionic gonadotropin {hCG} test with a minimum sensitivity of 25 international units per liter {IU/L} or equivalent units of beta-hCG {or hCG}]. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug)
5. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
6. Evidence of disease that may influence the outcome of the study within 4 weeks of the participants first planned dose; example, disorders of the gastrointestinal (GI) tract especially peptic ulceration, GI bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome, liver, kidney, chronic respiratory system, dermatological system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism. Participants with Gilbert's Syndrome are not allowed
7. Any history of GI or abdominal surgery or conditions that may affect absorption, metabolism or excretion of E7386 example, intestinal resections, hepatectomy, nephrectomy, digestive organ resection, fistulas or physiological/mechanical GI obstruction at screening
8. Contraindications to SmartPill^TM use: history of gastric bezoar, swallowing disorders, suspected or known strictures, severe dysphagia to food or pills, Crohn's disease or diverticulitis
9. Presence of non-removable metal objects such as metal plates, screws, etc, in the abdominal region of the body. Very small metal items (example, sterilization clips, hernia repair staples) are permitted
10. Acute diarrhea or constipation in the 7 days before the predicted Day 1. If screening occurs greater than (>) 7 days before the Day 1, this criterion will be determined on Day 1. Diarrhea will be defined as the passage of liquid feces and/or a stool frequency of >3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
11. Any abnormal clinical symptom or organ impairment found by medical history at screening, and physical examinations, clinical laboratory tests and vital signs
12. Hemoglobin, total white cell count, neutrophils or platelets below the lower limit of normal at screening. Alanine aminotransferase (ALT) >1.2*upper limit of normal (ULN) that is, up to 60 IU/L (men) and 42 IU/L (women) at screening
13. A prolonged QT/corrected QT (QTc) interval (corrected QT interval by Fridericia's formula [QTcF] >450 millisecond [msec]) as demonstrated by a repeated electrocardiogram at screening or baseline or a history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
14. Known history of clinically significant drug or food allergies or presently experiencing any seasonal or perennial allergy at screening
15. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results at screening
16. History of drug or alcohol dependency or abuse within the 2 years before screening, or those who have a positive urine drug test or breath alcohol test at screening or admission
17. Alcohol consumption in males >21 units per week and females >14 units per week (1 unit=1/2 pint beer, or a 25 milliliter (mL) shot of 40 percent (%) spirit, 1.5 to 2 units=125 mL glass of wine, depending on type)
18. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of >10 parts per million (ppm) at screening or admission
19. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
20. Currently enrolled in another clinical study or used any investigational drug or device within the 90 days prior to Day 1 or Period 1
21. Participants who are, or are immediate family members of, a study site or sponsor employee
22. Participants who do not have suitable veins for multiple venipunctures/cannulation as assessed by the investigator or delegate at screening
23. Receipt of blood products within 4 weeks of dosing, or donation of blood or plasma within the previous 3 months or loss of >400 mL of blood
24. Use of recreational drugs is prohibited
25. Use of any prescription drugs/herbal remedies or over-the-counter medications within 4 weeks or 14 days, respectively, before dosing (other than occasional use of up to 4 gram of paracetamol per day)
26. Any history of or concomitant medical condition that in the opinion of the investigator would compromise the participants ability to safely complete the study
27. Any lifetime history of psychiatric disease (including but not limited to depression or other mood disorders, bipolar disorder, psychotic disorders, including schizophrenia, panic attacks, anxiety disorders [if ever treated with medication]). The absence of a history of psychiatric disease should be documented by a checklist in the electronic case report form
28. Any lifetime suicidal behavior or ideation (per the Suicidal Behavior section of the Columbia-Suicide Severity Rating Scale [C-SSRS]) at screening
29. History or ongoing psychiatric disorder or psychiatric symptoms as evaluated by a physician at screening. Whenever possible, medical records should be reviewed to determine any history of psychiatric disorder or use of medications to treat psychiatric disorders
30. Evidence of current corona virus disease (COVID) 19 infection or ongoing/unrecovered sequelae COVID-19
31. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for E7386 | Day 1: 0-48 hours post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E7386 | Day 1: 0-48 hours post-dose
AUC (0-t): Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for E7386 | Day 1: 0-48 hours post-dose
AUC (0-inf): Area Under the Concentration-time Curve From Zero (Pre-dose) Extrapolated to Infinite Time for E7386 | Day 1: 0-48 hours post-dose
T1/2: Terminal Elimination Phase Half-life for E7386 | Day 1: 0-48 hours post-dose
CL/F: Apparent Total Clearance Following Extravascular Administration for E7386 | Day 1: 0-48 hours post-dose
Vz/F: Apparent Volume of Distribution at Terminal Phase for E7386 | Day 1: 0-48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.